CLINICAL TRIAL: NCT06503172
Title: The Clinical Effectiveness of Taiwanese Whole Grain Job's Tear on Muscle Health, Blood Glucose and Lipid Levels- a Randomized Controlled Trial
Brief Title: Whole Grain Job's Tear, Muscle Health, Blood Glucose and Lipid Level
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Taichung District Agricultural Research and Extension Station, Ministry of Agriculture, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04-005C
Record Dates: First submitted 2024-06-21; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Frailty; Hyperglycemia; Hyperlipidemia
MeSH Terms: conditions — Sarcopenia; Frailty; Hyperglycemia; Hyperlipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Taiwanese whole grain job's tear (Red job's tear) (Experimental): Taiwanese whole grain job's tear (Red job's tear)
  Interventions: Biological: Taiwanese whole grain job's tear (red job's tear)
- White job's tear (Active Comparator): White job's tear
  Interventions: Biological: White job's tear
- Active comparator group (Active Comparator): Active comparator group
  * serve as comparator group from week 0 to week 8,
  * assigned to red job's tear or white job's tear group from week 8 to week 16
  Interventions: Biological: Taiwanese whole grain job's tear (red job's tear); Biological: White job's tear

INTERVENTIONS:
Biological: Taiwanese whole grain job's tear (red job's tear) — 300cc drink made from red job's tear, 2 bottle/day from week 0 to week 8
  Arms: Active comparator group; Taiwanese whole grain job's tear (Red job's tear)
Biological: White job's tear — 300cc drink made from white job's tear, 2 bottle/day from week 0 to week 8
  Arms: Active comparator group; White job's tear

SUMMARY:
Background: This investigation aims to explore efficacy of Taiwanese whole grain job's tear on muscle health and blood glucose and lipid levels in community-dwelling older adults.

Methods: An open-label, 16-week, randomized controlled, cross-over trial involving participants with subject complaint of slower gait or weakness or fall in last year were recruited. The intervention group consumed Taiwanese whole grain job's tear (red job's tear) or white job's tear. Assessments included laboratory tests, functional assessments, and body composition.

ELIGIBILITY:
Inclusion Criteria:

People who aged 60-95 years

Patients with following characteristics:

feeling loss in activity detecting decline in self's walking speed. feeling tired of doing everything. having fall event in last year. People willing to follow the program and cooperate with us for following tracking.

People who are neither vegan nor vegetarian People agree and be able to sign the informed consent.

Exclusion Criteria:

People with any disease affecting their limbs, including:

having fracture on limbs in the past 6 months having severe arthritis in the past 6 months any other whom PI recognized as weak control of their nervous system( e.g.: Parkinson's disease and stroke).

People with intermittent limp caused by peripheral artery diseases People with weak control of mental disorder People with weak control of Cardiopulmonary disease People with weak control of Malignant tumor People with weak control of kidney diseases (eGFR <60ml/min/1.73) People with Visual impairment and Hearing disorder which cannot help to complete the program.

People who have underwent hormone treatment and planned to undergo hormone treatment during program session.

Any other condition that PI recognized as not suitable

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes of appendicular skeletal muscle index(ASMI) | 0, 8, 16 week
  ASMI=appendicular skeletal muscle mass(kg)/(height(m)2)
Changes of handgrip strength | 0, 8, 16 week
  Maximal handgrip strength of dominant hand (kg)
Changes of gait speed | 0, 8, 16 week
  Usual gait speed measured by 6-meter walking (m/s)
Changes of time required to finish timed up and go(TUG) test | 0, 8, 16 week
  Changes of time required to finish timed up and go(TUG) test

SECONDARY OUTCOMES:
Changes of inflammation marker | 0, 8, 16 week
  defined by hsCRP
Changes of insulin resistance | 0, 8, 16 week
  Measured by HOMA-IR
Changes of LDL | 0, 8, 16 week
  Changes of LDL
Changes of muscle biomarker 1 | 0, 8 week
  Measured by serum myostatin
Changes of muscle biomarker 2 | 0, 8 week
  Measured by serum follistatin
Changes of muscle biomarker 3 | 0, 8 week
  Measured by serum activin A

CONTACTS AND LOCATIONS:
Overall Officials: Anchun Hwang, Doctor, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No